CLINICAL TRIAL: NCT03022019
Title: Autologous Cell Suspension Grafting Using ReNovaCell in Non-segmental Vitiligo Patients: a Randomized Controlled Study
Brief Title: ReNovaCell in Non-segmental Vitiligo
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Futility
Sponsor: Netherlands Institute for Pigment Disorders (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); Avita Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: NL57683.018.16
Record Dates: First submitted 2017-01-12; First posted 2017-01-16 (Estimated); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Non-segmental Vitiligo; Vitiligo
Keywords: autologous cell suspension grafting; vitiligo; non-segmental; ReNovaCell
MeSH Terms: conditions — Vitiligo

ARMS (2):
- No ReNovaCell treatment (No Intervention): Lesion on the same patient that receives only standard therapy, no ReNovaCell treatment.
- ReNovaCell treatment (Experimental): Lesion on the same patient that receives the ReNovaCell treatment
  Interventions: Device: ReNovaCell

INTERVENTIONS:
Device: ReNovaCell
  Other Names: Autologous cell suspension grafting
  Arms: ReNovaCell treatment

SUMMARY:
Rationale:

Autologous epidermal cell suspension grafting is an effective method of surgical treatment in vitiligo, which is suitable for treating large areas with good cosmetic results. The RenovaCell Autologous Cell Harvesting Device (Avita Medical Europe Limited, Cambridge, UK) (previous name: ReCell) is a device which, compared to other forms of autologous epidermal cell suspension grafting, is easier in use showing similar results. Efficacy and safety of the ReCell device was proven in segmental vitiligo and piebaldism. However, the efficacy in non-segmental vitiligo is not yet confirmed in randomized controlled trials. The investigators hypothesize that grafting using the ReNovaCell device in combination with standard of care is also effective in stable non-segmental vitiligo and more effective than standard of care alone.

Objective:

Primary: to assess the efficacy and safety of ReNovaCell grafting combined with 311 nm UVB therapy and topical anti-inflammatory therapy for the treatment of stable non-segmental vitiligo. Secondary: to assess, satisfaction, cosmetic acceptability, noticeability and persistence of repigmentation after ReNovaCell transplantation.

Study design: Prospective, observer-blinded, randomised, within subject, controlled, study.

Study population: 20 patients ≥ 18 years with stable non-segmental vitiligo receiving standard of care (311 nm UVB therapy and topical anti-inflammatory therapy) for at least 6 months at the Netherlands Institute for Pigment Disorders (NIPD) at the Academic Medical Centre, University of Amsterdam.

Intervention: In patients already receiving standard of care (311 nm UVB therapy + topical anti-inflammatory therapy) 2 comparable depigmented regions are randomised to receive ReNovaCell grafting or no grafting. Standard of care will be given according to the standard treatment protocol of our institute.

Main study parameters/endpoints:

Primary outcome:

Objective assessment of the degree of repigmentation three and six months after ReNovaCell grafting with a digital image analysis system. To assess the pigmentation, the contours of pigmentation are copied on a transparent sheet before, three and six months after treatment, after which the sheets are scanned and digital image analysis is used to compute the affected surface. By comparing pre- and post-treatment pictures, the relative surface showing repigmentation expressed as percentage of the selected treated patch is computed.

Secondary outcomes:

* Patient Reported Outcomes: satisfaction, cosmetic acceptability, noticeability
* General patient assessed outcome per treatment region on a scale from 0-3 (poor, moderate, good or excellent).
* Visual assessment of percentage repigmentation by blinded observer and color match to normal skin
* Visual assessment of side effects per treatment region (hyperpigmentation, hypopigmentation and scarring on a scale from 0-3) by a blinded investigator.
* A small amount of the suspension of the included patients and the redundant lesional punchgrafts of all patients will be used for flow cytometric analyses of the cellular composition of the grafted cell suspension, and expression analysis of melanin synthesis-related genes. These data will be correlated to the clinical data.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: As the study involves large depigmented lesions, which are too large to treat in regular surgical treatment (punch grafting), patients will not miss any regular treatment. The time investment for the patient will be approximately 20 minutes for the punchgrafting session, 75 minutes for the cell suspension grafting session and 15 minutes for the three follow-up visits. Two of the five visits are part of the standard of care UVB follow-up regimen and are therefore not additional due to the study. Infection in the grafted area or the donor site may occur but is very rare; the risk of mild textural changes in the donor site is moderate. Hyperpigmentation of the treated area does occur often, although this improves over time in most cases. In case of improvement of the depigmentation, patients may receive another treatment for the (contralateral) untreated side.

ELIGIBILITY:
Inclusion Criteria:

* Patients with, non-segmental vitiligo receiving 6 months of standard of care, consisting of topical corticosteroids or immune modulators and NB-UVB phototherapy
* Age ≥18
* Patient is willing and able to give written informed consent
* At least two comparable (in location and diameter) depigmented lesions of at least 10 cm2 or one large lesion of at least 30 cm2 on the extremities, face or trunk.

Exclusion Criteria:

* Patients with signs of activity (spreading of lesions and/or koebnerisation) during standard of care treatment or showing depigmentation in the test punch grafting
* Skin type I
* Recurrent HSV skin infections
* Hypertrophic scars
* Keloid
* Cardiac insufficiency
* Patients with a history of hypersensitivity to (UVB or UVA) light and/or allergy to local anaesthesia.
* Patients who are pregnant or breast-feeding
* Patients not competent to understand what the procedures involves
* Patients with a personal history of melanoma or non-melanoma skin cancer
* Patients with atypical nevi.
* Known allergy to clarithromycin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-05-14 (Actual); Study Completion 2019-05-14 (Actual)

PRIMARY OUTCOMES:
degree of repigmentation | 3 and 6 months
  Objective assessment of the degree of repigmentation three and six months after ReNovaCell grafting with a digital image analysis system.

OTHER OUTCOMES:
Patient Reported Outcomes: satisfaction, cosmetic acceptability, noticeability | 6 months
Visual assessment of percentage repigmentation by blinded observer and color match to normal skin | 6 months
Visual assessment of side effects per treatment region | 6 months
  Visual assessment of side effects per treatment region (hyperpigmentation, hypopigmentation and scarring on a scale from 0-3) by a blinded investigator
flow cytometric analyses of the cellular composition of the grafted cell suspension | at time of autologous cell suspension grafting

CONTACTS AND LOCATIONS:
Locations (1):
- Nipd / Amc, Amsterdam, Netherlands